CLINICAL TRIAL: NCT03503773
Title: A Phase 2, Multicenter, Blinded, Sham Procedure-Controlled Trial of Renal Denervation by the Peregrine System Kit, in Subjects With Hypertension, in the Absence of Antihypertensive Medications
Brief Title: The TARGET BP OFF-MED Trial
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ablative Solutions, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR0014
Record Dates: First submitted 2018-03-23; First posted 2018-04-20 (Actual); Results first posted 2024-10-04 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Hypertension; Hypertension,Essential
Keywords: Renal Denervation; Neurolysis
MeSH Terms: conditions — Hypertension; Essential Hypertension | interventions — Ethanol

STUDY DESIGN:
Intervention Model Description: Subjects who continue to be eligible at the end of the run-in period will be randomized in a 1:1 ratio to one of the following 2 groups via central randomization (stratified by study site):
  * Treatment Arm: renal denervation (using the Peregrine Kit) performed with alcohol infused through the Peregrine Catheter
  * Sham Control Arm: only renal angiography performed
Who Masked: Participant, Outcomes Assessor
Masking Description: Blinded (The subject, sponsor, and hypertensionist/nephrologist performing the screening and follow-up assessments are blinded. The interventionalist and cath lab staff are unblinded.)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Arm: (Experimental): Renal denervation (using the Peregrine Kit) performed with alcohol infused through the Peregrine Catheter
  Interventions: Drug: Alcohol
- Sham Control Arm (Sham Comparator): Only renal angiography performed
  Interventions: Other: Sham control

INTERVENTIONS:
Drug: Alcohol — Alcohol is directly infused/delivered to the adventitial and periadventitial space of the renal arteries
  Arms: Treatment Arm:
Other: Sham control — endovascular, renal angiography
  Arms: Sham Control Arm

SUMMARY:
To obtain an assessment of the efficacy and safety of renal denervation by alcohol-mediated neurolysis using the Peregrine Kit in hypertensive subjects in the absence of antihypertensive medications.

ELIGIBILITY:
Inclusion Criteria:

1. Has 3 office blood pressure measurements with a mean office systolic blood pressure (SBP) of ≥140 mmHg and ≤180 mmHg, AND a mean office diastolic blood pressure (DBP) of ≥90 mmHg.
2. Subject is willing to discontinue any current antihypertensive medications during the run-in period and the post-treatment period.
3. Has a mean 24-hour ambulatory SBP of ≥135 mmHg and ≤170 mmHg with ≥70% valid readings

Exclusion Criteria:

1. Subject has renal artery anatomy abnormalities.
2. Subject has an estimated glomerular filtration rate (eGFR) of ≤45 mL/min/1.73 m2, based on the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation; or is on chronic renal replacement therapy.
3. Subject has documented sleep apnea.
4. Subject has any of the following conditions: severe cardiac valve stenosis, heart failure (New York Heart Association [NYHA] Class III or IV), chronic atrial fibrillation, and known primary pulmonary hypertension (>60 mmHg pulmonary artery or right ventricular systolic pressure).
5. Subject is pregnant or lactating at the time of enrollment or planning to become pregnant during the trial time period (female subjects only).
6. Subject is being treated chronically (e.g. daily use) with NSAIDs, immunosuppressive medications, or immunosuppressive doses of steroids. Aspirin therapy and nasal pulmonary inhalants are allowed.
7. Subject has a history of myocardial infarction, unstable angina pectoris, or stroke/TIA within 6 months prior to the planned procedure.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Actual)
Dates: Start 2018-09-24 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2024-01-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Felix Mahfoud, Prof.Dr.med., Principal Investigator — Universitätsklinikum des Saarlandes Klinik für Innere Medizin III Kardiologie, Angiologie und Internistische Intensivmedizin, Germany; Atul Pathak, Prof., Principal Investigator — Clinique Pasteur Hi-LAB, Toulouse, France
Locations (4):
- Cliniques Universitaires Saint-Luc, Brussels, Belgium
- Clinique Pasteur Toulouse, Toulouse, France
- Universitätsklinikum des Saarlandes, Homburg/Saar, Germany
- NIHR Barts Cardiovascular Biomedical Research Unit, London, United Kingdom

REFERENCES:
- [Background] Pathak A, Rudolph UM, Saxena M, Zeller T, Muller-Ehmsen J, Lipsic E, Schmieder RE, Sievert H, Halbach M, Sharif F, Parise H, Fischell TA, Weber MA, Kandzari DE, Mahfoud F. Alcohol-mediated renal denervation in patients with hypertension in the absence of antihypertensive medications. EuroIntervention. 2023 Sep 18;19(7):602-611. doi: 10.4244/EIJ-D-23-00088. PMID 37427416
- [Derived] Bertog S, Sharma A, Mahfoud F, Pathak A, Schmieder RE, Sievert K, Papademetriou V, Weber MA, Haratani N, Lobo MD, Saxena M, Kandzari DE, Fischell TA, Sievert H. Alcohol-Mediated Renal Sympathetic Neurolysis for the Treatment of Hypertension: The Peregrine Infusion Catheter. Cardiovasc Revasc Med. 2021 Mar;24:77-86. doi: 10.1016/j.carrev.2020.09.003. Epub 2020 Sep 7. PMID 32958438

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Enrolled and consented (n=350)
Period: Overall Study
Arm/Group | Sham Control Arm | Treatment Arm:
Started | 56 | 50
Completed | 44 (Completed 12-month follow-up and included in per-protocol population) | 43 (Completed 12-month follow-up and included in per-protocol population)
Not Completed | 12 | 7
Not completed — Not receiving bilateral treatment or an unsuccessful procedure | 0 | 2
Not completed — Receiving antihypertensive medications prior to evaluation of the primary ABPM | 8 | 4
Not completed — Not completing the primary ABPM | 3 | 1
Not completed — Not meeting inclusion/exclusion criteria | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment Arm: | Sham Control Arm | Total
Number analyzed (Participants) | 50 | 56 | 106
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.8 (11.0) | 54.4 (11.5) | 54.1 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 18 | 28
  Male | 40 | 38 | 78
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Belgium | 1 | 1 | 2
  United Kingdom | 7 | 9 | 16
  France | 7 | 6 | 13
  Germany | 28 | 30 | 58
  Netherlands | 4 | 4 | 8
  Ireland | 2 | 2 | 4
  United States | 1 | 4 | 5
eGFR [Mean (Standard Deviation); unit: mL/min per 1.73 m^2] | 85.8 (14.0) | 85.9 (13.0) | 85.8 (13.4)
Diabetes (type 2) [Count of Participants; unit: Participants] | 2 | 5 | 7
Smoking (current) [Count of Participants; unit: Participants] | 8 | 3 | 11
Peripheral vascular occlusive disease [Count of Participants; unit: Participants] | 1 | 1 | 2
Angiographically determined coronary artery disease [Count of Participants; unit: Participants] | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Changes in Systolic Ambulatory Blood Pressure
Description: Change from baseline in mean 24-hour ambulatory systolic blood pressure
Time Frame: Baseline to 8 weeks post-treatment
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Sham Control Arm | Treatment Arm:
Number analyzed (Participants) | 52 | 48
mmHg | -1.4 (8.6) | -2.9 (7.4)
Statistical Analysis 1: Comparison: Sham Control Arm vs Treatment Arm:; The null hypothesis to be tested is that there is no difference in the change in 24 hour mean SBP between treatment and sham control. The Type I error rate for rejecting the null hypothesis will be set at an alpha level of 0.05; Test type: Superiority; p = 0.2682, ANCOVA; Mean Difference (Final Values) = -1.5, 95% CI 2-sided [-4.8 to 1.7] — There was no formal hypothesis testing conducted in the study. 95% CIs are intended to be descriptive in nature only

2. Secondary Outcome: Change in Mean 24-Hour Ambulatory Systolic Blood Pressure at 6 Months
Description: Change from baseline in mean 24-hour ambulatory systolic blood pressure from baseline to 6 months
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Sham Control Arm | Treatment Arm:
Number analyzed (Participants) | 48 | 45
mmHg
  Mean 24-Hour Ambulatory Systolic Blood Pressure | 135.1 (11.7) | 134.1 (11.6)
  Change from baseline in Mean 24-Hour Ambulatory Systolic Blood Pressure | -13.4 (12.9) | -13.9 (11.6)
Statistical Analysis 1: Comparison: Sham Control Arm vs Treatment Arm:; Difference between treatment arms; Test type: Superiority; p = 0.6964, ANCOVA

3. Secondary Outcome: Change in Mean 24-Hour Ambulatory Systolic Blood Pressure at 12 Months
Description: Change from baseline in mean 24-hour systolic blood pressure at 12 months post-procedure
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Sham Control Arm | Treatment Arm:
Number analyzed (Participants) | 44 | 41
mmHg
  Mean 24-hour SBP | 133.7 (11.3) | 137.6 (11.4)
  Change from baseline in mean 24-hour SBP | -15.9 (13.1) | -10.6 (11.5)
Statistical Analysis 1: Comparison: Sham Control Arm vs Treatment Arm:; Between group difference; Test type: Superiority; p = 0.0775, ANCOVA

4. Secondary Outcome: Change in Office SBP at 8 Weeks
Description: Change from Baseline in mean office SBP to Week 8
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Sham Control Arm | Treatment Arm:
Number analyzed (Participants) | 54 | 50
mmHg
  Office SBP | 160.6 (16.3) | 155.4 (14.3)
  Change from Baseline in mean office SBP | 0.63 (13.24) | -4.0 (12.6)

5. Secondary Outcome: Change in Mean 24-Hour Ambulatory Diastolic Blood Pressure at 8 Weeks
Description: Change from baseline in mean 24-hour ambulatory diastolic blood pressure and 8 weeks post-procedure
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Sham Control Arm | Treatment Arm:
Number analyzed (Participants) | 55 | 50
mmHg
  Mean 24-hour ambulatory diastolic blood pressure | 91.0 (6.8) | 92.2 (7.6)
  Change from baseline in Mean 24-hour ambulatory diastolic blood pressure | -1.1 (6.6) | -2.0 (5.1)
Statistical Analysis 1: Comparison: Sham Control Arm vs Treatment Arm:; Between group difference; Test type: Superiority; p = 0.4734, ANCOVA

6. Secondary Outcome: Change in Mean 24-Hour Ambulatory Diastolic Blood Pressure at 6 Months
Description: Change from baseline in mean 24-hour ambulatory diastolic blood pressure at 6 months post-procedure
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Sham Control Arm | Treatment Arm:
Number analyzed (Participants) | 48 | 45
mmHg
  Mean 24-hour ambulatory diastolic blood pressure | 83.4 (9.0) | 83.0 (8.4)
  Change from baseline in Mean 24-hour ambulatory diastolic blood pressure | -8.0 (8.5) | -9.3 (6.9)

7. Secondary Outcome: Change in Mean 24-Hour Ambulatory Diastolic Blood Pressure at 12 Months
Description: Change from baseline in mean 24-hour diastolic blood pressure 12 months post-procedure
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Sham Control Arm | Treatment Arm:
Number analyzed (Participants) | 44 | 41
mmHg
  Mean 24-hour ambulatory diastolic blood pressure | 81.0 (7.9) | 85.6 (8.7)
  Change from baseline in Mean 24-hour ambulatory diastolic blood pressure | -9.8 (8.3) | -7.3 (7.5)
Statistical Analysis 1: Comparison: Sham Control Arm vs Treatment Arm:; Test type: Superiority; p = 0.0341, ANCOVA

8. Secondary Outcome: Number of Participants With Major Adverse Events (MAEs)
Description: Number of participants with major adverse events (MAEs) 30 days post-procedure
Time Frame: 30 days post procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Sham Control Arm | Treatment Arm:
Number analyzed (Participants) | 56 | 50
Participants | 1 | 1

9. Secondary Outcome: Use of Antihypertensive Medication(s)
Description: Use of antihypertensive medication at 8 weeks
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: medications
Arm/Group | Sham Control Arm | Treatment Arm:
Number analyzed (Participants) | 56 | 50
medications | 0.089 (0.288) | 0.060 (0.240)
Statistical Analysis 1: Comparison: Sham Control Arm vs Treatment Arm:; Test type: Superiority; p = 0.573, Fisher Exact; Mean Difference (Final Values) = -0.029, 95% CI 2-sided [-0.132 to 0.073]

10. Secondary Outcome: Change in Mean Daytime Ambulatory Systolic Blood Pressure at 8 Weeks
Description: Change from Baseline in Mean Daytime Ambulatory Systolic Blood Pressure to 8 Weeks
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Sham Control Arm | Treatment Arm:
Number analyzed (Participants) | 52 | 49
mmHg
  Mean Daytime Ambulatory Systolic Blood Pressure | 153.2 (12.0) | 150.6 (10.5)
  Change from Baseline in Mean Daytime Ambulatory Systolic Blood Pressure | -1.7 (9.9) | -3.2 (9.5)

11. Secondary Outcome: Change in Mean Daytime Ambulatory Systolic Blood Pressure at 6 Months
Description: Change from Baseline in Mean Daytime Ambulatory Systolic Blood Pressure to 6 Months
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Sham Control Arm | Treatment Arm:
Number analyzed (Participants) | 46 | 44
mmHg
  Mean Daytime Ambulatory Systolic Blood Pressur | 140.6 (12.3) | 139.7 (12.8)
  Change from Baseline in Mean Daytime Ambulatory Systolic Blood Pressure to 6 Months | -14.5 (13.7) | -14.0 (13.3)

12. Secondary Outcome: Change in Mean Daytime Ambulatory Systolic Blood Pressure at 12 Months
Description: Change from Baseline in Mean Daytime Ambulatory Systolic Blood Pressure to 12 Months
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Sham Control Arm | Treatment Arm:
Number analyzed (Participants) | 44 | 41
mmHg
  Mean Daytime Ambulatory Systolic Blood Pressure | 140.1 (12.1) | 143.5 (12.6)
  Change from Baseline in Mean Daytime Ambulatory Systolic Blood Pressure | -15.5 (13.6) | -10.5 (12.8)

13. Secondary Outcome: Mean Daytime Ambulatory Diastolic Blood Pressure
Description: Change from Baseline in Mean Daytime Ambulatory Diastolic Blood Pressure to 8 Weeks
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Sham Control Arm | Treatment Arm:
Number analyzed (Participants) | 54 | 50
mmHg
  Mean Daytime Ambulatory Diastolic Blood Pressure | 94.7 (9.7) | 95.2 (7.5)
  hange from Baseline in Mean Daytime Ambulatory Diastolic Blood Pressure | -1.4 (6.8) | -2.3 (6.8)

14. Secondary Outcome: Change in Mean Daytime Ambulatory Diastolic Blood Pressure at 6 Months
Description: Change from Baseline in Mean Daytime Ambulatory Diastolic Blood Pressure to 6 months
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Sham Control Arm | Treatment Arm:
Number analyzed (Participants) | 47 | 44
mmHg
  Mean Daytime Ambulatory Diastolic Blood Pressure | 87.6 (9.0) | 87.8 (9.2)
  Change from Baseline in Mean Daytime Ambulatory Diastolic Blood Pressure | -8.9 (8.6) | -9.3 (8.9)

15. Secondary Outcome: Change in Mean Daytime Ambulatory Diastolic Blood Pressure at 12 Months
Description: Change from Baseline in Mean Daytime Ambulatory Diastolic Blood Pressure to 12 Months
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Sham Control Arm | Treatment Arm:
Number analyzed (Participants) | 44 | 41
mmHg
  Mean Daytime Ambulatory Diastolic Blood Pressure | 86.0 (8.7) | 90.4 (9.6)
  Change from Baseline in Mean Daytime Ambulatory Diastolic Blood Pressure | -9.5 (8.7) | -7.6 (8.9)

16. Secondary Outcome: Change in Mean Nighttime Ambulatory Systolic Blood Pressure at 8 Weeks
Description: Change from Baseline in Mean Nighttime Ambulatory Systolic Blood Pressure to 8 Weeks
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Sham Control Arm | Treatment Arm:
Number analyzed (Participants) | 52 | 48
mmHg
  Mean Nighttime Ambulatory Systolic Blood Pressure | 136.9 (14.6) | 134.4 (11.6)
  Change from Baseline in Mean Nighttime Ambulatory Systolic Blood Pressure | -0.58 (12.17) | -3.3 (9.4)

17. Secondary Outcome: Change in Mean Nighttime Ambulatory Systolic Blood Pressure at 6 Months
Description: Change from Baseline in Mean Nighttime Ambulatory Systolic Blood Pressure to 6 Months
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Sham Control Arm | Treatment Arm:
Number analyzed (Participants) | 45 | 44
mmHg
  Mean Nighttime Ambulatory Systolic Blood Pressure | 125.6 (13.9) | 125.4 (12.1)
  Change from Baseline in Mean Nighttime Ambulatory Systolic Blood Pressure | -12.8 (14.1) | -13.4 (12.7)

18. Secondary Outcome: Change in Mean Nighttime Ambulatory Systolic Blood Pressure to 12 Months
Description: Change from Baseline in Mean Nighttime Ambulatory Systolic Blood Pressure to 12 Months
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Sham Control Arm | Treatment Arm:
Number analyzed (Participants) | 44 | 39
mmHg
  Mean Nighttime Ambulatory Systolic Blood Pressure | 123.1 (12.3) | 127.8 (10.7)
  Change from Baseline in Mean Nighttime Ambulatory Systolic Blood Pressure | -17.1 (14.4) | -11.8 (12.2)

19. Secondary Outcome: Change in Mean Nighttime Ambulatory Diastolic Blood Pressure at 8 Weeks
Description: Change from Baseline in Mean Nighttime Ambulatory Diastolic Blood Pressure to 8 weeks
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Sham Control Arm | Treatment Arm:
Number analyzed (Participants) | 52 | 48
mmHg
  Mean Nighttime Ambulatory Diastolic Blood Pressure | 82.5 (12.4) | 81.5 (8.4)
  Change from Baseline in Mean Nighttime Ambulatory Diastolic Blood Pressure | -0.44 (10.17) | -2.5 (7.3)

20. Secondary Outcome: Change in Mean Nighttime Ambulatory Diastolic Blood Pressure at 6 Months
Description: Change from Baseline in Mean Nighttime Ambulatory Diastolic Blood Pressure to 6 Months
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Sham Control Arm | Treatment Arm:
Number analyzed (Participants) | 46 | 45
mmHg
  Mean Nighttime Ambulatory Diastolic Blood Pressure | 75.8 (10.8) | 75.5 (9.2)
  Change from Baseline in Mean Nighttime Ambulatory Diastolic Blood Pressure | -7.4 (10.4) | -9.0 (8.0)

21. Secondary Outcome: Change in Mean Nighttime Ambulatory Diastolic Blood Pressure at 12 Months
Description: Change from Baseline in Mean Nighttime Ambulatory Diastolic Blood Pressure to 12 Months
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Sham Control Arm | Treatment Arm:
Number analyzed (Participants) | 44 | 39
mmHg
  Mean Nighttime Ambulatory Diastolic Blood Pressure | 72.8 (8.2) | 77.4 (7.8)
  Change from Baseline in Mean Nighttime Ambulatory Diastolic Blood Pressure | -10.8 (9.7) | -7.6 (8.1)

22. Secondary Outcome: Change in Mean Office SBP at 6 Months
Description: Change from Baseline in mean office SBP to 6 Months
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Sham Control Arm | Treatment Arm:
Number analyzed (Participants) | 51 | 45
mmHg
  mean office SBP | 145.7 (14.3) | 146.1 (16.4)
  Change from Baseline in mean office SBP to 6 Months | -14.7 (15.7) | -12.9 (15.6)

23. Secondary Outcome: Change in Mean Office SBP to 12 Months
Description: Change from Baseline in mean office SBP to 12 Months
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Sham Control Arm | Treatment Arm:
Number analyzed (Participants) | 50 | 41
mmHg
  mean office SBP | 147.8 (15.1) | 147.9 (18.5)
  Change from Baseline in mean office SBP to 12 Months | -13.2 (16.6) | -11.0 (15.3)

24. Secondary Outcome: Change in Mean Office DBP to 8 Weeks
Description: Change from Baseline in mean office DBP to 8 Weeks
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Sham Control Arm | Treatment Arm:
Number analyzed (Participants) | 54 | 50
mmHg
  mean office DBP | 97.3 (10.9) | 97.0 (9.4)
  Change from Baseline in mean office DBP to 8 Weeks | -1.1 (8.8) | -3.5 (7.6)

25. Secondary Outcome: Change in Mean Office DBP to 6 Months
Description: Change from Baseline in mean office DBP to 6 Months
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Sham Control Arm | Treatment Arm:
Number analyzed (Participants) | 51 | 45
mmHg
  mean office DBP | 89.7 (10.5) | 90.4 (9.4)
  Change from Baseline in mean office DBP to 6 Months | -8.4 (9.5) | -10.0 (9.0)

26. Secondary Outcome: Change in Mean Office DBP at 12 Months
Description: Change from Baseline in mean office DBP to 12 Months
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Sham Control Arm | Treatment Arm:
Number analyzed (Participants) | 50 | 41
mmHg
  mean office DBP | 88.5 (11.5) | 91.0 (11.0)
  Change from Baseline in mean office DBP to 12 Months | -9.6 (11.0) | -9.4 (9.4)

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Sham Control Arm | Treatment Arm:
All-Cause Mortality (participants affected / at risk) | 0/56 | 0/50
Serious Adverse Events (participants affected / at risk) | 9/56 | 7/50
Other Adverse Events (participants affected / at risk) | 42/56 | 41/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sham Control Arm (N=56) | Treatment Arm: (N=50)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 2 (2)
Abdominal abscess (Infections and infestations) | 0 (0) | 1 (1)
Appendicitis perforated (Infections and infestations) | 0 (0) | 1 (1)
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Haemoglobin decreased (Investigations) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Lumbar vertebral fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Sciatica (Nervous system disorders) | 1 (1) | 0 (0)
Urethral stenosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Lung neoplasm malignant (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Mitral valve repair (Surgical and medical procedures) | 1 (1) | 0 (0)
Aneurysm (Vascular disorders) | 0 (0) | 1 (1)
Haematoma (Vascular disorders) | 0 (0) | 1 (1)
Hypertensive crisis (Vascular disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sham Control Arm (N=56) | Treatment Arm: (N=50)
Oedema peripheral (General disorders) | 3 (3) | 1 (1)
Nasopharyngitis (Infections and infestations) | 4 (4) | 2 (2)
Post procedural haematoma (Injury, poisoning and procedural complications) | 4 (4) | 6 (6)
Blood pressure increased (Investigations) | 3 (3) | 2 (2)
Glomerular filtration rate decreased (Investigations) | 5 (5) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 2 (2)
Headache (Nervous system disorders) | 7 (7) | 11 (11)
Hypertension (Vascular disorders) | 5 (5) | 3 (3)
Hypertensive crisis (Vascular disorders) | 3 (3) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Chest discomfort (Cardiac disorders) | 0 (0) | 1 (1)
Dyspnoea exertional (Cardiac disorders) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 2 (2) | 1 (1)
Ocular discomfort (Eye disorders) | 0 (0) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1)
Coeliac artery compression syndrome (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastroenteritis viral (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haemorrhoids thrombosed (Gastrointestinal disorders) | 1 (1) | 0 (0)
Adverse drug reaction (General disorders) | 0 (0) | 1 (1)
Asthenia (General disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1)
Drug intolerance (General disorders) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1)
Oedema (General disorders) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 3 (3)
Peripheral swelling (General disorders) | 0 (0) | 1 (1)
Puncture site haematoma (General disorders) | 0 (0) | 1 (1)
Puncture site haemorrhage (General disorders) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Abdominal abscess (Infections and infestations) | 0 (0) | 1 (1)
Acute sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Appendicitis perforated (Infections and infestations) | 0 (0) | 1 (1)
Asymptomatic COVID-19 (Infections and infestations) | 1 (1) | 1 (1)
COVID-19 (Infections and infestations) | 2 (2) | 1 (1)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Sinusitis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Upper respiratory tract infection (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Arterial intramural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Joint injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post procedural complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Scratch (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Blood pressure diastolic increased (Investigations) | 0 (0) | 1 (1)
Blood sodium decreased (Investigations) | 0 (0) | 1 (1)
Glycosylated haemoglobin increased (Investigations) | 0 (0) | 1 (1)
Haemoglobin decreased (Investigations) | 1 (1) | 0 (0)
Gout (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Protein deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Joint effusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Lumbar vertebral fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Ageusia (Nervous system disorders) | 1 (1) | 0 (0)
Balance disorder (Nervous system disorders) | 1 (1) | 0 (0)
Disturbance in attention (Nervous system disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 2 (2)
Dizziness postural (Nervous system disorders) | 1 (1) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Multiple sclerosis (Nervous system disorders) | 1 (1) | 0 (0)
Restlessness (Nervous system disorders) | 0 (0) | 1 (1)
Sciatica (Nervous system disorders) | 1 (1) | 0 (0)
Sleep disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Nocturia (Renal and urinary disorders) | 1 (1) | 0 (0)
Nocturia (Renal and urinary disorders) | 0 (0) | 2 (2)
Urethral stenosis (Psychiatric disorders) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1)
Menopausal symptoms (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Lung neoplasm malignant (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Acarodermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Nail discolouration (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Apicectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Mitral valve repair (Surgical and medical procedures) | 1 (1) | 0 (0)
Varicose vein operation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Aneurysm (Vascular disorders) | 0 (0) | 1 (1)
Arterial disorder (Vascular disorders) | 0 (0) | 1 (1)
Dizziness (Vascular disorders) | 2 (2) | 1 (1)
Haematoma (Vascular disorders) | 2 (2) | 5 (5)
Hypertensive urgency (Vascular disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Peripheral artery occlusion (Vascular disorders) | 0 (0) | 1 (1)
Peripheral venous disease (Vascular disorders) | 0 (0) | 1 (1)
Post procedural haematoma (Vascular disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Vascular disorders) | 1 (1) | 0 (0)
Renal artery dissection (Vascular disorders) | 0 (0) | 1 (1)
Syncope (Vascular disorders) | 1 (1) | 0 (0)
Thrombophlebitis superficial (Vascular disorders) | 1 (1) | 0 (0)
Varicose vein (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-12-14): https://cdn.clinicaltrials.gov/large-docs/73/NCT03503773/Prot_000.pdf
  • Statistical Analysis Plan (2021-11-19): https://cdn.clinicaltrials.gov/large-docs/73/NCT03503773/SAP_001.pdf